CLINICAL TRIAL: NCT04748237
Title: Randomized Evaluation of Coronary Computed Tomographic Angiography in Intermediate-risk Patients Presenting to the Emergency Department With Chest Pain
Brief Title: Coronary Computed Tomographic Angiography in Intermediate-risk Chest Pain Patients
Acronym: FAST-CCTA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Dr. Tomas Jernberg, Principal Investigator, Clinical Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: KIDS2020-1
Record Dates: First submitted 2021-01-29; First posted 2021-02-10 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Chest Pain; Acute Coronary Syndrome; Coronary Artery Disease
MeSH Terms: conditions — Chest Pain; Acute Coronary Syndrome; Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Patients presenting to the ED with chest pain or other symptoms suggestive of ACS, without acute MI but with an intermediate risk (HEART-score >3) will after written informed consent be randomized to either a strategy with an initial coronary computed tomographic angiography or not.
Who Masked: Outcomes Assessor
Masking Description: Before adjudication, all documents will be masked regarding previous coronary computed tomographic angiography.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coronary computed tomopraphic angiography (Experimental): Patients randomized to strategy including early CCTA will receive standard care according to responsible physician and referred to a CCTA as soon as possible, preferably within 24 hours, but not later than within 21 days. Local scanning protocols can be used on ≥64-slice multi-detector CT scanners able to perform ECG-gated coronary angiography.
  The coronary angiography will be classified as normal (or near normal) or as having atherosclerosis (CAD). The report will also classify each vessel (left main, prox LAD, mid or distal LAD, LCX and RCA regarding degree of stenosis (no stenosis, 0-49%, ≥50%, or not possible to estimate because of calcification or technical reason).
  The result will be presented to the responsible physician as soon as possible and who will plan further care of the patients.
  Interventions: Diagnostic Test: Coronary computed tomopraphic angiography
- No Coronary computed tomopraphic angiography (No Intervention): Patients randomized to a strategy not including early CCTA will receive further care (including examinations) according to responsible physician but not include early CCTA. These patients will often undergo a non-invasive functional test, such as Exercise-ECG, stress echocardiography or nuclear imaging according to local routines, but not always.
  Regardless of diagnostic strategy, the responsible physician is encouraged to initiate secondary prevention measures if the investigations indicate signs of CAD, including medication with aspirin and statins.

INTERVENTIONS:
Diagnostic Test: Coronary computed tomopraphic angiography — CCTA as soon as possible, preferably within 24 hours, but not later than within 21 days.
  Arms: Coronary computed tomopraphic angiography

SUMMARY:
The aim is to determine whether a diagnostic strategy including early coronary computed tomographic angiography in intermediate-risk patients presenting to the Emergency Department with chest pain reduces the composite endpoint of death, readmission because of myocardial infarction or unstable angina requiring revascularization.

DETAILED DESCRIPTION:
Patients presenting to the ED with chest pain or other symptoms suggestive of ACS, without acute MI but with an intermediate risk (HEART-score >3) will after written informed consent be randomized to either a strategy with an initial CCTA or not.

Patients randomized to strategy including early CCTA will receive standard care according to responsible physician and perform a CCTA as soon as possible (in most cases within 24 hours, but at least within 21 days).The result will be presented to the responsible physician who will plan further care of the patients.

Patients randomized to a strategy not including early CCTA will receive further care (including examinations) according to responsible physician but not include early CCTA. These patients will often undergo a non-invasive functional test, such as Exercise-ECG, stress echocardiography or nuclear imaging according to local routines, but not always.

All patients should receive optimal prevention according to current guidelines. The responsible physician will be encouraged to initiate secondary prevention measures if examinations show signs of CAD.

The primary endpoint is composite of death, readmission because of MI or unstable angina requiring revascularization.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years.
2. Within 24 hours from presenting to the ED with chest pain or other symptoms suggestive of coronary artery disease (CAD)
3. HEART-score >3 (according to http://www.heartscore.nl/)
4. Written informed consent obtained

Exclusion Criteria:

1. Any condition that may influence the patient's ability to comply with study protocol.
2. Acute MI
3. Known obstructive CAD (>50%) or previous PCI or CABG.
4. Clear alternative diagnosis
5. Estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73m2
6. Major allergy to iodinated contrast media
7. Circumstances making high quality images unlikely.
8. Not a Swedish resident with a personal ID-number.
9. Pregnancy or breast feeding
10. Further investigation for CAD not indicated, due to limited life expectancy, quality of life or functional status
11. Previous inclusion in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2021-01-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The composite of death, readmission because of MI or unstable angina requiring revascularization | through study completion, an average of 5 year
  death of any cause, readmission because of MI (I21) or revascularization because of unstable angina not related to the index event

SECONDARY OUTCOMES:
Death or readmission because MI | through study completion, an average of 5 year
  death of any cause, readmission because of MI (I21)
Death | through study completion, an average of 5 year
  death of any cause
Cardiovascular death | through study completion, an average of 5 year
  death because of cardiovascular cause (I00-99)
MI (fatal or non-fatal) | through study completion, an average of 5 year
  readmission because of MI or death because of MI (I21)
Readmission because of unstable angina requiring revascularization | through study completion, an average of 5 year
  revascularization because of unstable angina not related to the index event.
Death, readmission because MI or stroke | through study completion, an average of 5 year
  death of any cause, readmission because of MI (I21) or stroke (I61-I64)
Stroke (fatal or non-fatal) | through study completion, an average of 5 year
  readmission because of stroke (I61-I64) or death because of stroke (I61-I64)
Resource use / Health care costs | through study completion, an average of 5 year
  Hospitalizations and investigations
Re-presentation to the ED because of chest pain | through study completion, an average of 5 year
  Re-presentation with chest pain as the main complaint
Invasive coronary angiography | through study completion, an average of 5 year
  Any invasive coronary angiography
Non-obstructive CAD at first invasive coronary angiography | through study completion, an average of 5 year
  Invasive coronary angiography without any significant stenoses
Angina | 1 year
  at least grade 1 according to Rose questionnaire
Use of prevention medications | 1, 2 and 3 years
  Use (dispensed prescriptions) of prevention medications (antiplatelet therapy, Statins, blood pressure lowering therapy)
Health-related quality of life | 1 year
  RAND-36: 8 domains/scales

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Jernberg, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Danderyd Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Other researchers can, after completion of study and the first report, apply for making analyses in collaboration with the steering group.